CLINICAL TRIAL: NCT01449097
Title: Comparison of the Efficacy of the Adductor-Canal-Blockade Versus the Femoral Nerve Block on Muscle Strength and Mobilization in Healthy Volunteers: a Randomized Study
Brief Title: Adductor-Canal-Blockade Versus the Femoral Nerve Block Effect on Muscle Strength and Mobilization in Healthy Volunteers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Pia Jaeger, Principal investigator, Rigshospitalet, Denmark
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SM2-PJ-11
Record Dates: First submitted 2011-10-06; First posted 2011-10-07 (Estimated); Last update posted 2011-12-22 (Estimated); Status verified 2011-12

CONDITIONS: Muscle Strength; Healthy Volunteers
Keywords: Adductor-Canal-blockade,; human volunteers,; US-guided nerve block; femoral nerve block

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Adductor-Canal-Blockade (Experimental)
  Interventions: Procedure: Adductor-Canal-Blockade
- The femoral nerve block (Active Comparator)
  Interventions: Procedure: The femoral nerve block
- Placebo (Placebo Comparator)
  Interventions: Procedure: Placebo

INTERVENTIONS:
Procedure: Adductor-Canal-Blockade — US-guided Adductor-Canal-blockade with Ropivacaine
  Arms: Adductor-Canal-Blockade
Procedure: The femoral nerve block — US-guided femoral nerve block with ropivacaine
  Arms: The femoral nerve block
Procedure: Placebo — US-guided Adductor-Canal-Blockade/femoral nerve block with saline
  Arms: Placebo

SUMMARY:
The aim of this study is to investigate the efficacy of the Adductor-Canal-Blockade versus the femoral nerve block versus placebo on muscle strength in healthy volunteers. The investigators hypothesize that the Adductor-Canal-Blockade results in a lesser reduction of the quadriceps muscle strength compared to the femoral nerve block.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* ASA 1
* BMI > 18 og < 25

Exclusion Criteria:

* Can not cooperate to the exam
* Do not speak or understand Danish
* Drug allergy
* Alcohol or drug abuse
* Daily consumption of analgetics on prescription
* Any drug intake within the last 48 hours
* Neuromuscular defects in the femoral nere, the obturator nerve or the muscles of the thigh.
* Previous surgery or trauma to the lower limb
* Diabetes Mellitus
* Intake of steroids, except steroids for inhalation
* Physical exercise within the last 24 hours prior to Day 1 and 2 of the study

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2011-10; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
the difference in quadriceps muscle strength between the Adductor-Canal-Blockade and placebo | 0-6 hours

SECONDARY OUTCOMES:
The difference in quadriceps muscle strength between the Adductor-Canal-Blockade and the femoral nerve block | 0-6 hours
The difference in quadriceps muscle strength between the placebo and the femoral nerve block | 0-6 hours
The difference in adductor muscle strength between the groups | 0-6 hours
The difference in mobilization between the groups | 0-6 hours

CONTACTS AND LOCATIONS:
Overall Officials: Pia Jæger, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Department of Anaesthesia, Centre of Head and Orthopaedics, Copenhagen University Hospital, Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Derived] Jaeger P, Nielsen ZJ, Henningsen MH, Hilsted KL, Mathiesen O, Dahl JB. Adductor canal block versus femoral nerve block and quadriceps strength: a randomized, double-blind, placebo-controlled, crossover study in healthy volunteers. Anesthesiology. 2013 Feb;118(2):409-15. doi: 10.1097/ALN.0b013e318279fa0b. PMID 23241723